CLINICAL TRIAL: NCT03771690
Title: A Replicated Crossover Study to Explore Individual Variability of Appetite Responses to a Standardised Meal and Any Moderating Influence of the FTO Gene
Brief Title: Individual Variability of Appetite Responses to a Standardised Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Teesside University (Other)
Responsible Party: Principal Investigator, Fernanda Reistenbach Goltz, Principal Investigator, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R17-P178
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Appetitive Behavior; Obesity; Genetic Predisposition to Disease
Keywords: Appetite; FTO; Ghrelin; Individual variability; Meal intake; Peptide YY
MeSH Terms: conditions — Appetitive Behavior; Obesity; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control 1 (No Intervention): After a 13 h overnight fast, participants will rest in the laboratory for the duration of the trial (09:00-11:00).
- Control 2 (No Intervention): After a 13 h overnight fast, participants will rest in the laboratory for the duration of the trial (09:00-11:00).
- Standardised meal 1 (Experimental): After a 13 h overnight fast, participants will rest in the laboratory for the duration of the trial (09:00-11:00). A standardised meal will be consumed at 10:00 which will provide 5025 kJ energy (47% carbohydrate, 9% protein, 44% fat).
  Interventions: Behavioral: Standardised meal
- Standardised meal 2 (Experimental): After a 13 h overnight fast, participants will rest in the laboratory for the duration of the trial (09:00-11:00). A standardised meal will be consumed at 10:00 which will provide 5025 kJ energy (47% carbohydrate, 9% protein, 44% fat).
  Interventions: Behavioral: Standardised meal

INTERVENTIONS:
Behavioral: Standardised meal — A standardised meal will be consumed at 10:00 which will provide 5025 kJ energy (47% carbohydrate, 9% protein, 44% fat).
  Arms: Standardised meal 1; Standardised meal 2

SUMMARY:
The aim of this study is to examine the interindividual variability of subjective and hormonal appetite responses to a standardised meal in healthy men and explore any moderating influence of the fat mass and obesity associated gene (FTO).

Participants homozygous for the obesity risk A allele (AA) or low risk T allele (TT) of FTO rs9939609 will complete two fasted control and two standardised meal (5025 kJ energy, 47% carbohydrate, 9% protein, 44% fat) conditions in randomised sequences. Ratings of perceived appetite and venous blood samples will be taken before and after the interventions. Interindividual differences in appetite responses and the potential moderating influence of the FTO gene will be examined using bivariate correlations and linear mixed modelling.

DETAILED DESCRIPTION:
Meal ingestion initiates a series of co-ordinated subjective and hormonal appetite responses. However, it is not known whether interindividual variability in appetite exists in response to a standardised meal. A recent approach proposed to quantify individual differences in the intervention response involves quantifying the participant-by-response interaction from replicated intervention and comparator arms. Using this approach (a replicated crossover study), the current study will (1) investigate whether the perceived appetite and appetite-related hormone responses to a standardised meal are reproducible on repeated occasions; (2) examine whether there is true individual variability in appetite responses to a standardised meal; and (3) determine whether the fat mass and obesity associated gene (FTO) moderates the magnitude of appetite responses to a standardised meal.

A total of 18 healthy men will be recruited according to their FTO rs9939609 genotype: 9 homozygous minor allele (AA) and 9 homozygous major allele (TT). Participants will complete four main experimental conditions each separated by an interval of at least three days: two fasted control and two standardised meal conditions. Participants will arrive at the laboratory at 09:00 after a 13 h overnight fast and a cannula will be inserted into an antecubital vein for blood sampling. After 60 min rest, a fasting venous blood sample and rating of perceived appetite will be taken (0 h; 10:00). Participants will rest throughout all four conditions but will be provided with a standardised breakfast meal after the fasting measurements during the two meal conditions. Breakfast will be consumed within 15 min and consist of croissants, butter, chocolate spread, cereal biscuits and milkshake which will provide 5025 kJ energy (47% carbohydrate, 9% protein, 44% fat). Subsequent venous blood samples will be taken at 0.5 h (10:30) and 1 h (11:00), and appetite perceptions will be assessed at 1 h (11:00).

Interindividual differences will be explored by correlating the two sets of response differences between meal and control conditions. Within-participant covariate-adjusted linear mixed models will be used to quantify participant-by-condition and FTO genotype-by-condition interactions.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous minor allele (AA) or major allele (TT) FTO rs9939609 genotype;
* Non-smoker;
* Weight stable for the previous 3 months.

Exclusion Criteria:

* Heterozygous FTO rs9939609 genotype (i.e., AT);
* Any medical conditions (e.g., diabetes, coagulation or bleeding disorders);
* Taking any medication that might influence appetite, fat metabolism or blood glucose;
* Dieting or restrained eating behaviours;
* Any food allergies.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Acylated ghrelin concentration | 1 hour (Plasma samples will be collected at 0 hour (pre) and 1 hour (post))
  Control adjusted pre-to-post change in plasma acylated ghrelin concentration

SECONDARY OUTCOMES:
Total peptide YY concentration | 1 hour (Plasma samples will be collected at 0 hour (pre) and 1 hour (post))
  Control adjusted pre-to-post change in plasma total peptide YY concentration
Insulin concentration | 0.5 hour (Plasma samples will be collected at 0 hour (pre) and 0.5 hour (post))
  Control adjusted pre-to-post change in plasma insulin concentration
Glucose concentration | 0.5 hour (Plasma samples will be collected at 0 hour (pre) and 0.5 hour (post))
  Control adjusted pre-to-post change in plasma glucose concentration
Rating of perceived hunger | 1 hour (Visual analogue scales will be completed at 0 hour (pre) and 1 hour (post))
  Control adjusted pre-to-post change in rating of perceived hunger. Perceived hunger will be measured using a 100 mm visual analogue scale anchored at 0, 'I am not hungry at all', and 100, 'I have never been more hungry'.
Rating of perceived satisfaction | 1 hour (Visual analogue scales will be completed at 0 hour (pre) and 1 hour (post))
  Control adjusted pre-to-post change in rating of perceived satisfaction. Perceived satisfaction will be measured using a 100 mm visual analogue scale anchored at 0, 'I am completely empty', and 100, 'I cannot eat another bite'.
Rating of perceived fullness | 1 hour (Visual analogue scales will be completed at 0 hour (pre) and 1 hour (post))
  Control adjusted pre-to-post change in rating of perceived fullness. Perceived fullness will be measured using a 100 mm visual analogue scale anchored at 0, 'Not full at all', and 100, 'Totally full'.
Rating of perceived prospective food consumption | 1 hour (Visual analogue scales will be completed at 0 hour (pre) and 1 hour (post))
  Control adjusted pre-to-post change in rating of perceived prospective food consumption. Perceived prospective food consumption will be measured using a 100 mm visual analogue scale anchored at 0, 'Nothing at all', and 100, 'A lot'.
  consumption

CONTACTS AND LOCATIONS:
Overall Officials: David Stensel, Principal Investigator — Loughborough University; Fernanda Reistenbach Goltz, Principal Investigator — Loughborough University; Greg Atkinson, Principal Investigator — Teesside University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goltz FR, Thackray AE, King JA, Dorling JL, Atkinson G, Stensel DJ. Interindividual Responses of Appetite to Acute Exercise: A Replicated Crossover Study. Med Sci Sports Exerc. 2018 Apr;50(4):758-768. doi: 10.1249/MSS.0000000000001504. PMID 29240652
- [Background] Atkinson G, Batterham AM. True and false interindividual differences in the physiological response to an intervention. Exp Physiol. 2015 Jun;100(6):577-88. doi: 10.1113/EP085070. Epub 2015 May 13. PMID 25823596
- [Background] Senn S, Rolfe K, Julious SA. Investigating variability in patient response to treatment--a case study from a replicate cross-over study. Stat Methods Med Res. 2011 Dec;20(6):657-66. doi: 10.1177/0962280210379174. Epub 2010 Aug 25. PMID 20739334
- [Background] Senn S. Mastering variation: variance components and personalised medicine. Stat Med. 2016 Mar 30;35(7):966-77. doi: 10.1002/sim.6739. Epub 2015 Sep 28. PMID 26415869
- [Derived] Goltz FR, Thackray AE, Atkinson G, Lolli L, King JA, Dorling JL, Dowejko M, Mastana S, Stensel DJ. True Interindividual Variability Exists in Postprandial Appetite Responses in Healthy Men But Is Not Moderated by the FTO Genotype. J Nutr. 2019 Jul 1;149(7):1159-1169. doi: 10.1093/jn/nxz062. PMID 31132105

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT03771690/SAP_000.pdf